CLINICAL TRIAL: NCT05327114
Title: Phase 2/3, Multistage, Multicenter, Randomized, Double-Blind, Placebo-Controlled Parallel Group Withdrawal Study to Evaluate the Efficacy and Safety of Nipocalimab Administered to Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: Efficacy and Safety Study of Nipocalimab for Adults With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109195; 80202135CDP3001 (Other: Janssen Research & Development, LLC); 2021-003234-37 (EudraCT Number); 2023-508425-28-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nipocalimab (Experimental): Participants in Stage A (Open-label) will receive a loading dose of nipocalimab (Dose 1) intravenous (IV) infusion on Day 1, followed by nipocalimab (Dose 2) IV infusion once every 2 weeks (q2w) from Week 2 to Week 12. Participants who demonstrate evidence of clinical improvement in Stage A (responders) will enter Stage B (Double-blind) and receive nipocalimab (Dose 2) IV infusion q2w starting on Day 1 up to Week 52. After completion of Stage B or discontinuation from Stage B due to relapse, participants will have the option to enter the open label extension (OLE) phase and receive nipocalimab (Dose 2) IV infusion q2w starting on OLE Day 1 until 2 years after marketing authorization in a participant's local country or until nipocalimab becomes available commercially or via other continued access program, whichever comes first.
  Interventions: Drug: Nipocalimab
- Placebo (Placebo Comparator): Participants receiving nipocalimab in Stage A and who demonstrate evidence of clinical improvement in Stage A (responders) will enter Stage B (Double-blind) and receive placebo IV infusion q2w starting on Day 1 up to Week 52. After completion of Stage B or discontinuation from Stage B due to relapse, participants will have the option to enter the open label extension (OLE) phase and receive nipocalimab (Dose 2) IV infusion q2w starting on OLE Day 1 until 2 years after marketing authorization in a participant's local country or until nipocalimab becomes available commercially or via other continued access program, whichever comes first.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nipocalimab — Nipocalimab will be administered intravenously.
  Other Names: JNJ-80202135; M281
  Arms: Nipocalimab
Drug: Placebo — Placebo will be administered intravenously.
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety and efficacy of nipocalimab compared to placebo in delaying relapse in adults with chronic inflammatory demyelinating polyneuropathy (CIDP) who initially respond to nipocalimab in Stage A.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (>=) 18 years of age at the time of consent and as applicable, must also meet the legal age of consent in the jurisdiction in which the study is taking place
* Diagnosed with Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) according to criteria of the European Academy of Neurology/Peripheral Nerve Society (EAN/PNS) 2021, progressing or relapsing forms. CIDP diagnosis to be adjudicated by independent committee during screening period
* Inflammatory Neuropathy Cause and Treatment (INCAT) disability score between 2 and 9 at the Run-In Baseline visit for participants entering Run-In, or Stage A Baseline visit for participants directly entering Stage A. Participants with an INCAT score of 2 at trial entry must have this score exclusively from the leg disability score
* Fulfilling any of the following treatment conditions: a) Currently treated with oral corticosteroids (CS) less than or equal to (<=) 20 milligrams (mg)/day; or b) Currently treated with pulsed CS, and/or intravenous immunoglobulin (IVIg) or subcutaneous immunoglobulin (SCIg) and the participant is willing to discontinue no later than the run-in baseline visit; or c) Currently treated with oral CS greater than (>) 20 mg/day and the participant is willing to taper to <=20 mg/day during the run-in period; or d) Without previous treatment (treatment naive); or treatment with CS and/or IVIg or SCIg discontinued at least 3 months prior to screening (untreated)
* Active disease as determined by CIDP Disease Activity Status (CDAS) score >= 3
* Other protocol-defined inclusion criteria will apply

Exclusion Criteria:

* Has a history of severe and/or uncontrolled hepatic (example, viral/alcoholic/autoimmune hepatitis/cirrhosis and/or metabolic liver disease), gastrointestinal, renal, pulmonary, cardiovascular, psychiatric, neurological or musculoskeletal disorder, hypertension and/or any other medical or uncontrolled autoimmune disorder(s) (example, diabetes mellitus) or clinically significant abnormalities in screening laboratory that, might interfere with the participants full participation in the study, or might jeopardize the safety of the participant or the validity of the study results
* Pure sensory CIDP or chronic immune sensory polyradiculopathy (CISP) (EAN/PNS definition)
* Any other disease that could better explain the participant's signs and symptoms, such as significant persisting neurological deficits from stroke or central nervous system (CNS) trauma or peripheral neuropathy from another cause such as connective tissue disease or systemic lupus erythematosus
* Polyneuropathy of other causes, including the following: Multifocal motor neuropathy (MMN); Monoclonal gammopathy of uncertain significance with antimyelin associated glycoprotein (anti-MAG) immunoglobulin M (IgM) antibodies; Hereditary motor neuropathy; Hereditary neuropathy with liability to pressure palsies (HNPP); Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin change syndromes; Lumbosacral radiculoplexus neuropathy; Polyneuropathy most likely due to diabetes mellitus; Polyneuropathy most likely due to systemic illnesses; Drug- or toxin-induced polyneuropathy Note: A concomitant polyneuropathy of other causes (example, a mild, stable diabetic polyneuropathy) is not necessarily exclusionary if chronic inflammatory demyelinating polyneuropathy (CIDP) is confirmed as the main diagnosis, as determined by the investigator and confirmed by the adjudication committee
* Has known allergies, hypersensitivity, or intolerance to nipocalimab or its excipients
* Other protocol-defined exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2027-05-14 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Stage B: Time to First Occurrence of a Relapse Event | Up to 52 weeks
  Stage B time to first occurrence of a relapse event will be reported.

SECONDARY OUTCOMES:
Stage A: Time to Initial Confirmed Evidence of Clinical Improvement (ECI) | 12 weeks
  Time to initial confirmed ECI will be reported.
Stage A: Percentage of Responders as Determined by ECI | 12 weeks
  Stage A percentage of responders as determined by ECI will be reported.
Stage A: Change from Baseline Over Time in Adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Scale Score | Baseline to 12 weeks
  Change from Stage A baseline over time in adjusted INCAT disability scale score will be reported. The INCAT disability scale is a clinician-rated assessment that measures activity limitation and degree of functional disability. The INCAT scale is an ordinal scale scored from 0 to 10, with higher scores indicating more disability.
Stage A: Change from Stage A Baseline Over Time in Medical Research Council (MRC) Muscle Grading Scale Sum Score | Baseline to 12 weeks
  Change from Stage A baseline over time in MRC muscle grading scale sum score will be reported. The MRC muscle grading scale is a clinician-rated outcome that provides a strength rating (on a scale from 0 [no visible contraction] to 5 [normal]) in 6 muscles collected bilaterally: deltoid, biceps, wrist extensors, iliopsoas, quadriceps, tibialis anterior. Lower scores indicate greater impairment.
Stage A: Change from Baseline Over Time in Inflammatory Rasch-Built Overall Disability Scale (I-RODS) Centile Score | Baseline to 12 weeks
  Change from Stage A baseline over time in I-RODS centile score will be reported. The I-RODS comprises of 24 items representing common daily activities that address upper and lower limb disability and range in difficulty from very easy to very difficult. Lower scores indicate greater activity and social participation limitations.
Stage A: Change from Baseline Over Time in Mean Grip Strength (Dominant Hand) | Baseline to 12 weeks
  Change from Stage A baseline over time in mean grip strength (dominant hand) will be reported. Grip Strength is a quantifiable, objective performance outcome measure of hand strength, which can be measured using various devices (for example, Martin Vigorimeter and Jamar Dynamometer).
Stage A: Change from Baseline Over Time in Mean Grip Strength (Non-Dominant Hand) | Baseline to 12 weeks
  Change from Stage A baseline over time in mean grip strength (non-dominant hand) will be reported. Grip Strength is a quantifiable, objective performance outcome measure of hand strength, which can be measured using various devices (for example, Martin Vigorimeter and Jamar Dynamometer).
Stage B: Time to First Adjusted INCAT Disability Scale Score Deterioration Relative to Baseline | Up to 52 weeks
  Time to first adjusted INCAT disability scale score deterioration relative to Stage B baseline will be reported.
Stage B: Time to First Switch to Intravenous Immunoglobulin (IVIg) or Other Standard of Care (SoC) as a Result of Investigator-assessed Lack of Efficacy as Confirmed by an Independent RAC Relative to Baseline | Up to 52 weeks
  Time to first switch to IVIg or other SoC as a result of investigator-assessed lack of efficacy as confirmed by an independent Relapse Adjudication Committee (RAC) relative to Stage B baseline will be reported.
Stage B: Change from Baseline Over Time in Adjusted INCAT Disability Score | Up to 52 weeks
  Change from Stage B baseline over time in adjusted INCAT disability score will be reported.
Stage B: Change from Baseline Over Time in MRC Muscle Grading Scale Sum Score | Up to 52 weeks
  Change from Stage B baseline over time in MRC Muscle Grading Scale Sum score will be reported.
Stage B: Change from Baseline Over Time in I-RODS Centile Score | Up to 52 weeks
  Change from Stage B baseline over time in I-RODS centile score will be reported.
Stage B: Change from Baseline Over Time in Mean Grip Strength (Dominant Hand) | Up to 52 weeks
  Change from Stage B baseline over time in mean grip strength (dominant hand) will be reported. Grip Strength is a quantifiable, objective performance outcome measure of hand strength, which can be measured using various devices (for example, Martin Vigorimeter and Jamar Dynamometer).
Stage B: Change from Baseline Over Time in Mean Grip Strength (Non-Dominant Hand) | Up to 52 weeks
  Change from Stage B baseline over time in mean grip strength (non-dominant hand) will be reported. Grip Strength is a quantifiable, objective performance outcome measure of hand strength, which can be measured using various devices (for example, Martin Vigorimeter and Jamar Dynamometer).
Stage B: Number of Participants with Binary Response Endpoint Satisfying all 4 Conditions: a) An Improved Adjusted INCAT Disability Score Compared to Baseline; b) Not Relapsing; c) Not Switching to SoC; d) Not Discontinuing Treatment | Up to 52 weeks
  Number of participants with Binary response endpoint satisfying all 4 conditions: a) an improved adjusted INCAT Disability Score compared to Stage B baseline; b) not relapsing; c) not switching to SoC; d) not discontinuing treatment, will be reported.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Stage A: 12 weeks; Stage B: Up to 52 weeks
  An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment
Percentage of Participants with Serious Adverse Events (SAEs) | Stage A: 12 weeks; Stage B: Up to 52 weeks
  SAE is an adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly/birth defect; suspected transmission of any infectious agent via a medicinal product or medically important.
Number of Participants with Change in Electrocardiogram (ECG) Values Over Time | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with change in ECG values over time will be reported.
Number of Participants with Change in Vital Signs Values Over Time | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with change in vital signs values over time will be reported.
Number of Participants with Change in Clinical Laboratory Values Over Time | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with change in clinical laboratory values over time will be reported.
Number of Participants with Clinically Significant ECG Abnormalities | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with clinically significant ECG abnormalities will be reported.
Number of Participants with Clinically Significant Vital Signs Abnormalities | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with clinically significant vital signs abnormalities will be reported.
Number of Participants with Clinically Significant Clinical Laboratory Abnormalities | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with clinically significant clinical laboratory abnormalities will be reported.
Percentage of Participants with Suicidal Ideation or Suicidal Behavior based on the Columbia-Suicide Severity Rating Scale (C-SSRS) | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Percentage of participants with suicidal ideation or suicidal behavior based on the C-SSRS will be reported.
Serum Nipocalimab Concentrations Over Time in Participants Receiving Active Study Intervention | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Serum nipocalimab concentrations over time in participants receiving active study intervention will be reported.
Number of Participants with Anti-drug Antibodies (ADA) to Nipocalimab | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with ADA to Nipocalimab will be reported.
Titers of ADA to Nipocalimab | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Titers of ADA to nipocalimab will be reported.
Number of Participants with Neutralizing Antibodies (NAb) to Nipocalimab | Stage A: 12 weeks; Stage B: Up to 52 weeks
  Number of participants with NAb to Nipocalimab will be reported.
Change from Baseline in Total Serum Immunoglobulin (IgG) Concentrations Levels Over Time | Stage A: Baseline to 12 weeks; Stage B: Baseline up to 52 weeks
  Change from baseline in total serum IgG concentrations levels over time will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (103):
- United States (13):
  - IMMUNOe Health and Research Centers, Centennial, Colorado
  - Healthcare Innovations Institute Inc, Coral Springs, Florida
  - Neurology Associates PA, Maitland, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Beaumont Hospital Royal Oak, Royal Oak, Michigan
  - The Neurological Institute of New York, New York, New York
  - South Shore Neurologic Associates - Patchogue, Patchogue, New York
  - The Neurological Institute, PA, Charlotte, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Austin Neuromuscular Center, Austin, Texas
  - Advocate Health - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Argentina (2):
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Gral Agudos Ignacio Pirovano, Buenos Aires
- Australia (2):
  - The Alfred Hospital, Melbourne
  - Gold Coast University Hospital, Parkwood
- China (18):
  - Peking University First Hospital, Beijing
  - Xuanwu Hospital ,Capital Medical University, Beijing
  - Beijing Tiantan Hospital, Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital of Central Sourth University, Changsha
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Chifeng Municipal Hospital, Chifeng
  - Fujian Medical University Union Hospital, Fuzhou
  - The First Affiliated Hospital Sun Yat sen University, Guangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Qianfoshan hospital of Shandong Province, Jinan
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Huashan Hospital Fudan University, Shanghai
  - Tong Ren Hospital Shanghai Jiao Tong University school of medicine, Shanghai
  - Tangdu hospital the Fourth Military Medical, Xi'an
  - Xi 'an GaoXin Hospital, Xi'an
- Colombia (2):
  - Fundación Cardiovascular de Colombia - Instituto del Corazón Floridablanca, Floridablanca
  - Instituto Neurológico de Colombia, Medellín
- Czechia (3):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Pardubicka krajska nemocnice a s, Pardubice
- France (6):
  - CHU Bordeaux, Bordeaux
  - Hospices Civils de Lyon HCL, Bron
  - Hopital de Bicetre, Le Kremlin-Bicêtre
  - Hopital PASTEUR, Nice
  - Hopital de la Pitie Salpetriere, Paris
  - CHRU Strasbourg, Strasbourg
- Germany (5):
  - Judisches Krankenhaus Berlin, Berlin
  - St. Josef-Hospital, Ruhr-Universität Bochum, Bochum
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Leipzig, Leipzig
  - St Josefs Krankenhaus Potsdam Sanssouci, Potsdam
- Greece (3):
  - Attikon General Hospital of Athens, Athens
  - Patras University Hospital, Pátrai
  - Papageorgiou General Hospital Of Thessaloniki, Thessaloniki
- Italy (4):
  - Azienda Ospedaliera Universitaria San Martino di Genova, Genova
  - Azienda Ospedaliera di Rilievo Nazionale A Cardarelli, Naples
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Japan (19):
  - National Hospital Organization Asahikawa Medical Center, Asahikawa
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - Tokai University Hospital, Isehara
  - Kobe City Medical Center General Hospital, Kobe
  - National Center of Neurology and Psychiatry, Kodaira-shi
  - Saitama Medical Center, Koshigaya
  - Kumamoto University Hospital, Kumamoto
  - Chubu Rosai Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - Kindai University Hospital, Osaka Sayama Shi
  - National Hospital Organization Sendai Medical Center, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga Gun
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - Tenri Hospital, Tenri
  - Ehime University Hospital, Toon-shi
  - Toyama University Hospital, Toyama
  - Yamaguchi University Hospital, Ube
- Mexico (2):
  - i Can Oncology Center, Monterrey
  - Clinical Research Institute S.C., Tlalnepantla
- Poland (4):
  - Centrum Medyczne, Chorzów
  - Specjalistyczne Gabinety Lekarskie, Krakow
  - Prywatny Gabinet Lekarski, Lublin
  - Clinical Research Center sp z o o MEDIC R s k, Poznan
- Portugal (3):
  - Hospital Garcia de Orta, Almada
  - Hospital de Braga, Braga
  - Centro Hospitalar de Sao Joao Epe, Porto
- South Korea (3):
  - Kyunghee University Medical Center, Seoul
  - Konkuk University Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hosp. Gral. Univ. de Alicante, Alicante
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Univ. de Basurto, Bilbao
  - Hosp. Univ. Donostia, Donostia / San Sebastian
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Virgen Macarena, Seville
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Shin Kong Wu Ho Su Memorial Hospital, Taipei
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Devon & Exeter Hospital, Devon
  - NHS Greater Glasgow and Clyde, Glasgow
  - Royal Free Hospital, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency